CLINICAL TRIAL: NCT01660139
Title: Use of Alternative Medicine Among Outpatients in Dermatology and Primary Care Clinics
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Maria Colavincenzo, Assistant Professor, Department of Dermatology, Northwestern University
Other Study IDs: STU67142
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Dermatologic Disorders
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dermatology Clinic Patients: Patient attending dermatology clinics
- Primary Clinic Patients: Patient attending primary care clinics

SUMMARY:
This study is to assess the practice of complementary and alternative medicine (CAM) for skin related conditions among patients in the Primary Care and Dermatology clinics.

DETAILED DESCRIPTION:
This study aims to determine the prevalence and characteristics complementary and alternative medicine (CAM) usage among Primary Care and Dermatology clinic patients through the use of an anonymous, self-completed written survey. This survey will assess the prevalence and regularity of CAM usage (with and without concurrent use of allopathic therapies), the reasons for CAM usage, perceived success with CAM usage, and socioeconomic status, in both Dermatology and Primary Care patients. We will then compare these elements of CAM usage between the two clinic patient populations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Presents for a clinic appointment with a dermatologist or primary care physician
* English-speaking

Exclusion Criteria:

* Less than 18 years or older
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending clinic appointments in dermatology and primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of complementary and alternative medicine usage among patients in the clinics | 5 minutes to complete survey
  At the clinic appointment, patients will be given a survey that asks about whether the patient uses complementary and alternative medicine for skin related issues.

SECONDARY OUTCOMES:
Characteristics of the patients complementary and alternative medicine use | 5 minutes to complete survey
  Patients who practice complementary and alternative medicine will be asked about what and how they practice their complementary and alternative medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Colavincenzo, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Result] Tindle HA, Davis RB, Phillips RS, Eisenberg DM. Trends in use of complementary and alternative medicine by US adults: 1997-2002. Altern Ther Health Med. 2005 Jan-Feb;11(1):42-9. PMID 15712765
- [Result] Parkman CA. CAM therapies and nursing competency. J Nurses Staff Dev. 2002 Mar-Apr;18(2):61-5; quiz 66-7. doi: 10.1097/00124645-200203000-00001. PMID 11984258
- [Result] Ernst E. The usage of complementary therapies by dermatological patients: a systematic review. Br J Dermatol. 2000 May;142(5):857-61. doi: 10.1046/j.1365-2133.2000.03463.x. PMID 10809840
- [Result] Ernst E, Pittler MH, Stevinson C. Complementary/alternative medicine in dermatology: evidence-assessed efficacy of two diseases and two treatments. Am J Clin Dermatol. 2002;3(5):341-8. doi: 10.2165/00128071-200203050-00006. PMID 12069640
- [Result] Smith N, Shin DB, Brauer JA, Mao J, Gelfand JM. Use of complementary and alternative medicine among adults with skin disease: results from a national survey. J Am Acad Dermatol. 2009 Mar;60(3):419-25. doi: 10.1016/j.jaad.2008.11.905. Epub 2009 Jan 20. PMID 19157642
- [Result] Fuhrmann T, Smith N, Tausk F. Use of complementary and alternative medicine among adults with skin disease: updated results from a national survey. J Am Acad Dermatol. 2010 Dec;63(6):1000-5. doi: 10.1016/j.jaad.2009.12.009. Epub 2010 Oct 8. PMID 20933300
- See also: Northwestern University Department of Dermatology Actively Enrolling Research Trials — http://www.feinberg.northwestern.edu/depts/dermatology/research/clinical-trials/ctu-active%20trials.htm